CLINICAL TRIAL: NCT00903981
Title: A Randomized, Placebo Controlled, Double Blind, Multicenter Therapeutic Confirmatory Clinical Study for the Evaluation of the Efficacy and Safety of Avanafil in the Patients With Erectile Dysfunction
Brief Title: Therapeutic Confirmatory Study to Evaluate the Efficacy and Safety of Avanafil
Acronym: ALERT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: ChoongWae Pharma Corporation(Hyun Yoon Jeong), ChoongWae Pharma Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CWP-AVA-301
Record Dates: First submitted 2009-05-18; First posted 2009-05-19 (Estimated); Last update posted 2010-04-23 (Estimated); Status verified 2009-02

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — avanafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Avanafil 100mg (Experimental)
  Interventions: Drug: Avanafil
- Avanafil 200mg (Experimental)
  Interventions: Drug: Avanafil
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Avanafil — 2 tablets(Avanafil 100mg tablet + Placebo 200mg tablet), 30 minutes before sexual intercourse
  Arms: Avanafil 100mg
Drug: Avanafil — 2 Tablets(Avanafil 200mg tablet + Placebo 100mg tablet), 30 minutes before sexual intercourse
  Arms: Avanafil 200mg
Drug: Placebo — 2 Tablets(Placebo 100mg tablet + Placebo 200mg tablet), 30 minutes before sexual intercourse
  Arms: Placebo

SUMMARY:
The purpose of this study is to confirm the efficacy and the safety of Avanafil 100mg, 200mg or placebo administered orally for 12 weeks in patients with erectile dysfunction. The efficacy is evaluated by IIEF, SEP Q2 and Q3 and GEAQ and the safety is evaluated by laboratory tests, vital signs, physical examination and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* male subjects aged 19 to 70 with history of erectile dysfunction for at least 6 months
* subjects have stable monogamous relationships
* their partners are free from pregnancy and lactation and well prevent conception
* subjects consented to participate in the clinical study in writing
* subjects attempted sexual intercourse at least 4 times in separate days during 4 weeks' free run-in period, and failure rate is over 50%

Exclusion Criteria:

* history of spinal cord injury or radical prostatectomy
* subjects whose penises are anatomically deformed
* erectile dysfunction due to neurogenic or endocrine cause
* subjects who have uncontrolled major psychiatric disorder and do not accept therapies or have significant neurological abnormalities
* history of cancer chemotherapy within 1 year
* subjects who are addicted to alcohol or have continuously misused dependent drugs
* subjects who have hepatic dysfunction(GOP,GPT ≥ 3xUNL) or renal dysfunctions(serum creatinine > 2.0)
* subjects who have uncontrollable diabetes(FPG>180)
* subjects sho have proliferative diabetic retinopathy
* history of stroke, transient ischemic attacks, myocardial infarction, heart failure that needs to be medically treated, unstable angina or fatal arrhythmia or coronary artery bypass graft within 6 months
* serious hypotension or uncontrollable severe hypertension
* hematological disorders that is likely to be developed into priapism such as sickle cell disease, multiple myeloma, leukemia
* subjects who have retinitis pigmentosa
* subjects who suffered from serious GI bleeding disorder within 1 year
* subjects who took other PDE5 inhibitors or ED therapies within 2 weeks
* subjects who use non-concomitant medications(Nitrate/NO donors, Androgens, anti-androgen, trazodone, Anticoagulant,over-the-counter drugs known to inhibit the activity of CYP3A4)
* history of hypersensitivity to the PDE5 inhibitors or not responded to them
* subjects who have hypoactive sexual desire
* subjects who have no intention of having sexual intercourses 4 times in separate days during 4 weeks' free run-in period
* subjects who took other investigational products within 30 days before this clinical study
* subjects who are judged to be unsuitable to the clinical study by other reasons

Ages: 19 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2009-03; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Change of EF domain score in the IIEF(The International Index of Erectile Function) | 12 weeks

SECONDARY OUTCOMES:
Change of successful rate in SEPQ2,Q3,Q4,Q5 Change of score in other domains of IIEF Change of IIEF Q3 and Q4 score GEAQ The rate of normal erectile function | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jong Kwan Park, PhD, Principal Investigator — Chonbuk National University Hospital; Se Woong Kim, PhD, Principal Investigator — Catholic Seoul medical center; Jae Suk Hyun, PhD, Principal Investigator — Gyeongsang National University Hospital; Je Jong Kim, PhD, Principal Investigator — Korea University; Nam Cheol Park, PhD, Principal Investigator — Pusan National University Hospital; Sung Won Lee, PhD, Principal Investigator — Samsung Medical Center; Jae Seung Paick, PhD, Principal Investigator — Seoul National University Hospital; Tae young Ahn, PhD, Principal Investigator — Asan Medical Center; Ki Hak Moon, PhD, Principal Investigator — Yeungnam University Hospital; Woo Sik Chung, PhD, Principal Investigator — Ewha womans university hospital; Kweon Sik Min, PhD, Principal Investigator — Inje university Pusan paick hospital; Jun Kyu Suh, PhD, Principal Investigator — Inha University Hospital; Kwang Sung Park, PhD, Principal Investigator — Chonnam National University Hospital; Dae Yul Yang, PhD, Principal Investigator — Kangdong Sacred Heart Hospital
Locations (1):
- Chonbuk national university hospital, Jeonju, Cholabukdo, South Korea